CLINICAL TRIAL: NCT04550767
Title: Bacterial Infections in People Who Inject Psychoactive Substances
Brief Title: : Bacterial Infections in Injecting Drug Users
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0523
Record Dates: First submitted 2020-09-03; First posted 2020-09-16 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Bacterial Infection
Keywords: Psychoactive substance; Intravenous substance abuse; Injection drug user; Risk reduction; Psychoactive substances
MeSH Terms: conditions — Bacterial Infections; Substance Abuse, Intravenous; Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- local infections: local infections
- systemic infections: systemic infections

SUMMARY:
Bacterial infections in people who inject psychoactive substances

DETAILED DESCRIPTION:
In context of an increase of bacterial infections in people who inject psychoactive substances (PS) all around the world and a lack of available scientific data, the investigators decided to set up a descriptive study on bacterial infection types and determinants in Injection Drug Users (IDUs).

Through a multidisciplinary approach between hospital departments (e.g. infectious diseases, emergency and addictology), the local addiction management and liaison team (ELSA) and the regional addictovigilance center, data were collected on appearance and course of bacterial infections in IDUs hospitalized at Montpellier University Hospital, France.

This study aims to provide medical data in order to better understand those infections and their determinants and provide information for potential future more specific observational studies.

The regional addictovigilance center is a member of the French Addictovigilance Network, which was established to monitor the potential for abuse and dependence of PS, and to provide information on the risk of addiction and advice for public health decision making, under the supervision of the French National Agency for Medicines and Health Products Safety. This surveillance system is principally based on spontaneous reporting by healthcare professionals and patients that is regulated by law. Collected data were extracted from those spontaneous reports (composed by data from the medical file*, DxCare or notification by medical team). First data were collected in 2012.

In addition, the investigators offered patients to fill in an anonymous questionnaire** on hygiene habits which was not mandatory and had no influence on treatment, and was offered during the ELSA team intervention (questions from the questionnaire are classical risk reduction question on injection and hygiene practices).

Main results are the description of the infections and injection practices. There is no control group per se as all included patients are IDUs and have a bacterial infection. But the investigators infection (such as abscess or skin and soft tissue) and those with a systemic infection. The two groups were established after the recruitment was completed. This comparative analysis is only performed in order to better understand the development of infections. Descriptive and comparative analyses was performed by the Department of Medical Information.

*Data collected :

* Age
* Sex
* Past history of bacterial infection linked to injection of a psychoactive substance
* HIV and HCV status
* Injected psychoactive substance
* Injection practices (frequency, route, location)
* Diagnosis
* Bacterial analysis
* Treatments and course

  * Hygiene questionnaire (attached file)

ELIGIBILITY:
Inclusion criteria:

* Bacterial infection occurring in injection drug users and linked to injection
* Hospitalized at Montpellier University Hospital

Exclusion criteria:

* No injection
* No use of a psychoactive substance
* Viral or fungal infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all injection drug users, hospitalized at Montpellier University Hospital for bacterial infection related to the injection of one or several psychoactive substance(s).
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Types of bacterial infections | 1 day
  Types of bacterial infections : local or systemic:
Psychoactive substances involved in each type of bacterial infections | 1 day
  Psychoactive substances involved in each type of bacterial infections
Types of injections in each type of infections | 1 day
  Types of injections in each type of infections

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Peyrière, PH, Study Director — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC